CLINICAL TRIAL: NCT05091437
Title: Doubling Outcomes by Lung Cancer Early Diagnosis: An Observational, Study to Collect Real-world Evidence (RWE) on the Management of Pulmonary Nodules Across Latin-America
Brief Title: DOuBLED - Doubling Outcomes by Lung Cancer Early Diagnosis
Acronym: DOuBLED
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: INCUNA (Scientific and Technical partner) (Unknown)
Responsible Party: Sponsor
Other Study IDs: D133FR00176
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Nodules
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- Retrospective: All eligible subjects with solid or subsolid (part solid, pure ground glass) lung nodule identified in the past; more preciously from March 2019 to the study initiation date. [ Fleischner Society 2017 guidelines for nodules size and definition (≥ 6 mm and < 3 cm) for subject inclusion].
  Interventions: Diagnostic Test: Observational study
- Prospective: All eligible subjects with solid or subsolid (part solid, pure ground glass) lung nodule identified in imaging exams in routine clinical practice, prior to 30 days of informed consent given [ Fleischner Society 2017 guidelines for nodules size and definition (≥ 6 mm and < 3 cm)) for subject inclusion]. Subjects identified from different sources (Nodules identified incidentally and in lung cancer screening programs) will be considered.
  Interventions: Diagnostic Test: Observational study

INTERVENTIONS:
Diagnostic Test: Observational study — Incidental lung nodules identification

SUMMARY:
Early diagnosis of LC in the asymptomatic stage through intentional screening programs and/or incidental pulmonary nodule identification and follow-up are known to improve outcomes significantly. There are large gaps in the screening and early detection of LC, especially in LMIC - driven by multifactorial aspects, including a variety of socioeconomic and infrastructural factors, mainly due to limitations in the required network of specialized human resources and technical capacity. Identifying LC at an early stage allows for treatment that is more likely to be curative, thereby improving survival.

The present study aims to characterize the lung nodule journey in different hospitals/clinics across Latin America, describing the use of health resources, time to diagnosis, stage at diagnosis, and time to treatment depending on the source of nodule identification in two different cohorts (retrospective and prospective).

DETAILED DESCRIPTION:
This non-interventional observational study will capture data (retrospective and prospective cohorts) from around 20 to 25 hospitals/clinics to report lung nodules (patients' journey) in Latin America.

Objectives and Hypotheses:

Primary objective

• To describe the lung nodule patient journey from the time of nodule identification through its final diagnosis, staging, and treatment decision.

Note: Lung nodules identified from different settings would be nodules identified incidentally and in lung cancer screening programs.

Secondary objective(s)

* To determine the medical specialties involved in the lung nodule study journey.
* To describe a medical specialist who first identifies the lung nodule (referral patterns).
* To estimate the proportion of benign and malignant nodules.
* To understand health care resource utilization from nodule detection to final diagnosis and management.
* Time from nodule identification until a final diagnosis and treatment decision.
* Treatment decision and specialties involved in the decision.

Study Population:

Adult ≥ 35 years of age with solid or subsolid (part solid, pure ground glass) lung nodules identified in different settings, including nodules identified incidentally and nodules identified in lung cancer screening programs could be targeted. The study population will comprise two cohorts, one prospective for subjects starting the study of pulmonary nodules since site activation and onwards, and other retrospective for subjects who started the study of pulmonary nodules from March 2019.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥ 35 years of age)

  * a) Prospective cohort: All eligible subjects with solid or subsolid (part solid, pure ground glass) lung nodule identified in imaging exams in routine clinical practice, prior to 30 days of informed consent given [please refer to: Fleischner Society 2017 guidelines for nodules size and definition (≥ 6 mm and < 3 cm)) for subject inclusion]. Subjects identified from different sources (Nodules identified incidentally and in lung cancer screening programs) will be considered OR b) Retrospective cohort: All eligible subjects with solid or subsolid (part solid, pure ground glass) lung nodule identified in the past; more preciously from March 2019 to the study initiation date. [Please refer to: Fleischner Society 2017 guidelines for nodules size and definition (≥ 6 mm and < 3 cm) for subject inclusion].
  * Written informed consent to have medical data collected and stored for the prospective cohort and as guided by the local regulations for the retrospective cohort..

Exclusion Criteria:

* Subjects unable to undergo any lung diagnostic procedure.

  * Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years or are deemed by the investigator to be at low risk for recurrence of that malignancy
  * Subjects with calcified lung nodules with an established diagnosis

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (older than 35 years) who meet inclusion and exclusion criteria will be selected from the participants hospitals/clinics
Sampling Method: Non-Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Time of nodule identification up to diagnosis and treatment | 24 months
  Description of the lung nodule patient journey from the time of nodule identification through its final diagnosis, staging, and treatment decision.

CONTACTS AND LOCATIONS:
Overall Officials: Larisa Ramirez, MD, Study Director — AstraZeneca
Locations (14):
- Research Site, CABA, Argentina
- Brazil (3):
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Chile (2):
  - Research Site, Antofagasta
  - Research Site, Concepción
- Colombia (2):
  - Research Site, Bogotá
  - Research Site, Cundinamarca
- Research Site, San José, Costa Rica
- Research Site, Santo Domingo, Dominican Republic
- Mexico (3):
  - Research Site, Monterrey, Nuevo León
  - Research Site, Estado de México
  - Research Site, Mexico City
- Research Site, Panama City, Panama

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133FR00176&attachmentIdentifier=93a78782-9089-44b5-9b19-8f52ef40adbc&fileName=DOuBLED_Clinical_Study_Report_(CSR)_Synopsis_F.pdf&versionIdentifier=